CLINICAL TRIAL: NCT01371318
Title: Wound EMR to Decrease Limb Amputations in Persons With Diabetes
Brief Title: Online Wound Electronic Medical Record (OWEMR) to Decrease Amputations in Diabetics
Acronym: OWEMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Warren, Principal Investigator, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HS019218-01 (AHRQ)
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Wounds; Diabetes Complications; Diabetic Foot; Foot Ulcer
Keywords: diabetic foot ulcer; amputation; wounds; diabetic foot; diabetes complications
MeSH Terms: conditions — Wounds and Injuries; Diabetes Complications; Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OWEMR (Experimental): Medical centers will be randomized to use the Online Wound Electronic Medical Record to enhance care of patients with diabetic foot ulcers
  Interventions: Other: Online Wound Electronic Medical Record
- Standard of Care (No Intervention): Medical/wound centers will be randomized to continue routine care of patients with diabetic foot ulcers

INTERVENTIONS:
Other: Online Wound Electronic Medical Record — Online Wound Electronic Medical Record is a medical informatics tool that synthesizes data about complex wound problems from multiple sources and is innovative in its capability to performing these critical tasks: i) identification of the information needed to make treatment decisions at the point of care in real time ii) use intelligent search and report features to identify patients who require emergency interventions, and iii) provide evidence-based clinical decision support to clinicians
  Arms: OWEMR

SUMMARY:
The purpose of this study is to determine whether using the OWEMR as part of the standard of care for Diabetic Foot Ulcers reduces the rate of lower limb amputations and to quantify the relationship between glycemic control and the rate of amputation secondary to chronic foot ulcers in Type II Diabetes.

DETAILED DESCRIPTION:
The Online Wound Electronic Medical Record (OWEMR) is a medical informatics tool that synthesizes data about complex wound problems from multiple sources and is innovative in its capability to performing these critical tasks: i) identification of the information needed to make treatment decisions at the point of care in real time ii) use intelligent search and report features to identify patients who require emergency interventions, and iii) provide evidence-based clinical decision support to clinicians. Use of the OWEMR includes digital photography as an objective measurement of wound healing rates.

ELIGIBILITY:
* Signed informed Consent
* Type I or II diabetes*
* A break in the skin on the foot ≥ 0.5cm2
* 18 yrs of age or older
* Hemoglobin A1c value within the last 120 days
* No use of Investigational Agents /Devices on study or within 30 days prior to enrollment
* Subjects who will be locally available for the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1609 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Lower extremity amputation secondary to diabetic foot ulcer | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Warren, MD, Principal Investigator — NYU School of Medicine
Locations (13):
- United States (13):
  - Phoenix VA Hospital, Phoenix, Arizona
  - University of Arizona, Tuscon, Arizona
  - Western University Health Sciences, Pomona, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - Aiyan Diabetes Center, Evans, Georgia
  - Elks Wound Center, Meridian, Idaho
  - Mayo Clinic, Rochester, Minnesota
  - North Shore Long Island Jewish Health System, Lake Success, New York
  - Bellevue Hospital, New York, New York
  - Metropolitan Hospital, New York, New York
  - Lincoln Hospital, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas